CLINICAL TRIAL: NCT04420234
Title: A Single-center Phase I Clinical Study Evaluating the Pharmacokinetics and Safety of Single and Multiple Oral Administration of Narfurine Hydrochloride Orally Disintegrating Tablets in Chinese Healthy Adult Subjects
Brief Title: A Pharmacokinetics and Safety Study of Narfurine Hydrochloride Orally Disintegrating Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSS-Remitch-HD-I-01
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-06

CONDITIONS: Improvement of Pruritus in Hemodialysis Patients
Keywords: narfurine hydrochloride orally disintegrating tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacokinetics study of single and multiple administration (Experimental): During the study session, 30 healthy subjects will be administered a single and multiple dose of narfurine hydrochloride orally disintegrating tablets 5 µg (2.5 µg/table) to evaluate the pharmacokinetic parameters and the safety profile.
  Interventions: Drug: narfurine hydrochloride orally disintegrating tablets

INTERVENTIONS:
Drug: narfurine hydrochloride orally disintegrating tablets — Subjects swallowed 2 tablets of test drug (2.5 µg/tablet) with saliva at about 8:00 AM on D1; swallowed 2 tablets of test drug (2.5 µg/tablet) with saliva at about 8:00 AM starting on D4. Dosing for 7 consecutive days (D10 last dose in the morning).

SUMMARY:
Main objective: To evaluate the pharmacokinetics of single and multiple oral administration of narfurine hydrochloride orally disintegrating tablets in Chinese healthy adult subjects.

Secondary objective: To evaluate the safety profile of single and multiple oral administration of narfurine hydrochloride orally disintegrating tablets in Chinese healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old <= age <= 40 years old, male or female;
2. Weight: male >= 50 kg, female >= 45 kg; body mass index (BMI) in the range of 19-26 kg / m2 (including 19 and 26);
3. Important indicators including physical examination, vital signs examination, electrocardiogram examination, laboratory examination, and chest X-ray examination are normal or within the acceptable range of the sponsors or researchers;
4. During the trial and within 3 months after the last medication, there is no parenting plan and reliable contraceptive measures could be taken;
5. Fully understand the purpose and requirements of this trial, voluntarily participate in clinical trials and sign a written informed consent form, and can complete the entire trial process according to the trial requirements.

Exclusion Criteria:

1. Those who are known to have a history of allergies, allergic diseases or allergies to the test preparation and any of its components or related preparations;
2. Those who have a clear medical history of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders or serious infections and serious injuries, or other diseases that are not suitable for participating in clinical trials (such as history of mental illness, etc.)
3. Those who have donated blood or lost blood >= 400mL within 3 months before enrollment;
4. Those who have taken any drugs (including prescription drugs and over-the-counter drugs), vitamins, and Chinese herbal medicines within 2 weeks before screening;
5. Those who have participated in clinical trials of other drugs or medical devices within 3 months before being selected;
6. Those who is or was a drug addict or positive in drug abuse screening test;
7. Those who is or was an alcoholic (drinking more than 14 standard units per week. 1 standard unit contains 14g alcohol, such as 360mL beer or 45mL spirits with 40% alcohol or 150mL wine), or positive in urine alcohol test.
8. Smokers or those with an average daily smoking volume of more than 5 cigarettes within 3 months before screening, and those with a positive nicotine test;
9. Those who is positive in Hepatitis B surface antigen (HBsAg), HCV antibody, Treponema pallidum antibody and HIV antibody;
10. Female subjects who are in the lactation period or is positive in the pregnancy test during the screening period or clinical trial;
11. Those who have used any drugs that is CYP3A4 inhibitor or inducer within 4 weeks before signing the informed consent form, see Appendix 3 for details;
12. People with long-term insomnia and those with the habit of taking sleeping pills;
13. People with habitual constipation;
14. Those who is diagnosed abnormal or with clinical significance in physical examination, vital signs examination, electrocardiogram or clinical laboratory examination, etc.,
15. Those who have undergone surgery that can affect the absorption, distribution, metabolism, excretion of drugs, or have any gastrointestinal diseases that may affect the absorption of drugs, or those who are determined by the investigator to be unsuitable for enrollment;
16. Those who consume excessive amounts of tea, coffee and / or caffeinated beverages (more than 8 cups, 1 cup = 250mL) every day within 30 days before screening
17. Those who took grapefruit or grapefruit juice and drinks or foods containing St. John's wort (hypericum perforatum), ginseng, ginkgo, valerian, and echinacea within 48 hours before administration;
18. Those who is diagnosed abnormal or have clinical significance by researchers in the chest X-ray examination;
19. Those who develop new diseases during the pre-study screening stage or before study medication;
20. Those who cannot tolerate venipuncture blood collection;
21. Those who are thought to be unsuitable for participating in the trial by the researchers because of other factors.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
AUC AUC | Day1 to Day13
  Area Under the Plasma Concentration-time Curve
Cmax | Day1 to Day13
  Maximum Observed Plasma Concentration
Tmax | Day1 to Day13
  Time to Reach the Maximum Plasma Concentration
t1/2 | Day1 to Day13
  Elimination half-life
Kel | Day1 to Day13
  Elimination rate constant
CL/F CL/F | Day1 to Day13
  Apparent clearance
Vd/F | Day1 to Day13
  Apparent distribution volume based on terminal elimination phase
MRT | Day1 to Day13
  Mean residence time
Css_max | Day1 to Day13
  Steady state peak concentration
Css_min | Day1 to Day13
  Steady state Valley concentration
Css_av | Day1 to Day13
  Steady state average concentration
DF | Day1 to Day13
  Volatility index
Safety and tolerance indicators | Day1 to Day13
  AE and SAE

CONTACTS AND LOCATIONS:
Overall Officials: jian liu, master, Principal Investigator — The First Affiliated Hospital,ZheJiang Univercity
Locations (1):
- The First Affiliated Hospital,ZheJiang Univercity, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No